CLINICAL TRIAL: NCT01943357
Title: Improving the Self Management Skills of Older Adults With Diabetes
Brief Title: Improving Self Management Skills of Older Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Principal Investigator, Kate Lorig, professor emertius, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 26679; 109554 (Other Grant/Funding Number: NCOA)
Record Dates: First submitted 2013-09-09; First posted 2013-09-16 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes; Diabetes
Keywords: diabetes; patient education; self management; health improvement
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetes Self-Management Program (Experimental): Behavioral: Diabetes Self Management Program. Consists of either a six-week small-group face-to-face program with two peer leaders or an six-week peer-facilitated Internet-based program.
  Interventions: Behavioral: Diabetes Self Management Program

INTERVENTIONS:
Behavioral: Diabetes Self Management Program — The interventions include modeling and action-planning to enhance self-efficacy.
  Other Names: Better Choices Better Health--Diabetes

SUMMARY:
The study will help determine if the Better Choices Better Health Diabetes program (community-based or online, also known as the Diabetes Self-Management Program) improves the hbA1C of people with Type-II diabetes. The investigators will also examine 1) symptoms (fatigue, sleep, low blood sugar symptoms, depression, shortness of breath), 2) healthy behaviors (blood sugar monitoring; taking medications as prescribed; getting eye, foot, kidney and cholesterol exams; and activity), 3) the use of health care services. This project is a translational study to demonstrate the effectiveness of the intervention in the context of a major insurer.

DETAILED DESCRIPTION:
Self-report questionnaires and hbA1c capillary blood collection kits will be administered at baseline (prior to the intervention), six-months and twelve-months. Differences between baseline and followup scores will be used to determine if participants have benefited from the intervention, using intent-to-treat methodology. Subgroups and delivery method (small-group or on-line) will be compared using repeated measures and analyses of covariance.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* WellPoint insurance or medicare supplement plan participant
* 18 years or older

Exclusion Criteria:

* Treatment for cancer in past year
* Pregnant
* Under 18
* Previously taken a Stanford self-management program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Metabolic control HbA1C | Baseline to 12 months

SECONDARY OUTCOMES:
Symptom:fatigue | Baseline to 12 months
  Single item visual numeric scale. Examined at baseline, 6 months and 12 months. Paired t-tests used to assess if change significant.
symptom: sleep | Baseline to 12 months
  Single item visual numeric scale. Examined at baseline, 6 months and 12 months. Paired t-tests used to assess if change significant.
symptom: PHQ-8 depression | Baseline to 12 months
  8-item scale. Examined at baseline, 6 months and 12 months. Paired t-tests used to assess if any changes are significant.
symptoms: hypoglycemic index | Baseline to 12 months
  7-item scale. Examined at baseline, 6 months and 12 months. Paired t-tests used to assess if any changes are significant.
health behavior: blood glucose monitoring | Baseline to 12 months
  Self report of how often monitor glucose at baseline, 6 months and 12 months. Paired t-tests used to assess if any changes are significant.
health behavior: medication adherence | baseline to 12 months
  3-item scale collected at baseline, 6 months and 12 months. Paired t-tests used to assess if any changes are significant.
Health behavior: communication with physician | baseline to 12 months
  3-item scale collected at baseline, 6 months and 12 months. Paired t-tests used to assess if any changes are significant.
health behavior: exercise | baseline to 12 months
  Minutes of exercise during last week self-reported at baseline, 6-months and 12-months. Paired t-tests used to assess if any changes are significant.
health behavior/utilization: frequency of exams | baseline to 12 months
  Self report of how often examine feet and have eye, cholesterol and kidney levels tested. Collected at baseline, 6 months and 12 months. Paired t-tests used to assess if any changes are significant.
Health care utilization | baseline to 12 months
  Physician, ED, hospital visits in last six-months. Self reported at baseline, 6 months and 12 months. Paired t-tests used to assess if any changes are significant.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lorig, DPH, Principal Investigator — Stanford School of Medicine
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States